CLINICAL TRIAL: NCT02373371
Title: Efficacy and Safety of Metvix® Natural Daylight Photodynamic Therapy Versus Conventional Metvix® Photodynamic Therapy in Subject With Mild Actinic Keratoses
Brief Title: Actinic Keratoses Treatment With Metvix® in Combination With Light
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I14034
Record Dates: First submitted 2015-02-16; First posted 2015-02-27 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2018-08

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — methyl 5-aminolevulinate; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daylight (Experimental): Metvix® (160mg/g) and Photodynamic Therapy Daylight One session at baseline
  Interventions: Drug: Metvix®; Procedure: Photodynamic Therapy Daylight
- Conventional treatment (Active Comparator): Metvix® (160mg/g) and Photodynamic Therapy Blue light One session at baseline
  Interventions: Drug: Metvix®; Procedure: Photodynamic Therapy Blue light

INTERVENTIONS:
Drug: Metvix®
Procedure: Photodynamic Therapy Blue light — Photodynamic therapy (PDT) is a medical treatment that utilizes a photosensitizing molecule (Metvix) and a blue light source to activate the applied drug
  Arms: Conventional treatment
Procedure: Photodynamic Therapy Daylight — Photodynamic therapy (PDT) is a medical treatment that utilizes a photosensitizing molecule (Metvix) and a the day light to activate the applied drug
  Arms: Daylight

SUMMARY:
The main objective of this study is to compare efficacy and safety of Metvix® natural daylight photodynamic therapy with those of Metvix® conventional photodynamic therapy in subjects with mild actinic keratoses (intra-individual comparison)

ELIGIBILITY:
Inclusion Criteria:

* Male or female above 18 years;
* Subject with clinical diagnosis of mild Actinic Keratosis (AK) on the face or the scalp with or without clinical diagnosis of moderate AK on the target areas (TAs);

Exclusion Criteria:

* Subject with clinical diagnosis of at least one severe AK on TAs
* Subject with clinical diagnosis of other skin disease (including non-melanoma skin cancer) on the TAs;
* Subject with pigmented AK on the TAs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges University Hospital, Limoges, France

REFERENCES:
- [Result] Assikar S, Labrunie A, Kerob D, Couraud A, Bedane C. Daylight photodynamic therapy with methyl aminolevulinate cream is as effective as conventional photodynamic therapy with blue light in the treatment of actinic keratosis: a controlled randomized intra-individual study. J Eur Acad Dermatol Venereol. 2020 Aug;34(8):1730-1735. doi: 10.1111/jdv.16208. Epub 2020 Feb 21. PMID 31955461

RESULTS

PARTICIPANT FLOW:
Groups:
- Daylight: Metvix® (160mg/g) and Photodynamic Therapy Daylight One session at baseline
  Metvix®
  Photodynamic Therapy Daylight: Photodynamic therapy (PDT) is a medical treatment that utilizes a photosensitizing molecule (Metvix) and a the day light to activate the applied drug
- Conventional Treatment: Metvix® (160mg/g) and Photodynamic Therapy Blue light One session at baseline
  Metvix®
  Photodynamic Therapy Blue light: Photodynamic therapy (PDT) is a medical treatment that utilizes a photosensitizing molecule (Metvix) and a blue light source to activate the applied drug
Period: Overall Study
Arm/Group | Daylight | Conventional Treatment
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daylight | Conventional Treatment | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Median (Inter-Quartile Range); unit: year] | 75.0 [67.0 to 83.0] | 75.0 [67.0 to 83.0] | 75.0 [67.0 to 83.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  France | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Number of Treated Mild Lesions Per Side at Week 12
Description: The number of lesions is assessed at baseline (before treatment) and 12 weeks later.
  The difference in lesions is recorded for each patient. The mean of disappeared lesions are then calculated for all patients.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Daylight | Conventional Treatment
Number analyzed (Participants) | 13 | 13
number of lesions | 19.6 (6.0) | 20.0 (6.9)
Statistical Analysis 1: Comparison: Daylight vs Conventional Treatment; Main analysis: * nbDPKAdispM3 the number of KA disappeared at M3 after treatment with DPDT compared to the inclusion layer, * nbCPKAdispM3 the number of KA disappeared at M3 after treatment with conventional blue light, The primary endpoint is: differenceM3 = nbDPKAdispM3 - nbCPKAdispM3 The main analysis will consist of a signed Wilcoxon rank test for matched data testing whether "difference M3" is significantly different from 0; Test type: Superiority; p = 0.8460, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pain Assesment
Description: Pain assesment with a VAS Pain scale
  Visual analog scale [VAS] is a continuous scale comprised of a horizontal scale of 10 cm length . The scale is anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10).
Time Frame: at inclusion (after treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daylight | Conventional Treatment
Number analyzed (Participants) | 13 | 13
units on a scale | 1.2 (1.9) | 5.1 (2.1)

3. Secondary Outcome: Lesions Disappearance Rate at 1 Months From Baseline.
Description: The number of lesions is assessed at baseline (before treatment) and 1 month later.
  The difference in lesions is recorded for each patient. The rate is the quotient: " difference in lesions between baseline and at 1 month "/nubmer of lesions at baseline
Time Frame: 0(baseline),1 month
Measure: Mean (Standard Deviation); unit: percentage of disappeared lesions
Arm/Group | Daylight | Conventional Treatment
Number analyzed (Participants) | 13 | 13
percentage of disappeared lesions | 89.6 (7.2) | 94.6 (4.8)
Statistical Analysis 1: Comparison: Daylight vs Conventional Treatment; Test type: Superiority; p = 0.0005, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Lesions Disappearance Rate at 6 Months From Baseline.
Description: The number of lesions is assessed at baseline (before treatment) and 6 month later.
  The difference in lesions is recorded for each patient. The rate is the quotient: " difference in lesions between baseline and at 6 month "/nubmer of lesions at baseline
Time Frame: 0(baseline), 6 month
Measure: Mean (Standard Deviation); unit: percentage of disappeared lesions
Arm/Group | Daylight | Conventional Treatment
Number analyzed (Participants) | 13 | 13
percentage of disappeared lesions | 90.9 (5.9) | 94.7 (5.4)
Statistical Analysis 1: Comparison: Daylight vs Conventional Treatment; Test type: Superiority; p = 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: which adverse event data were collected over 6 months
Arm/Group | Daylight | Conventional Treatment
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daylight (N=13) | Conventional Treatment (N=13)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes